CLINICAL TRIAL: NCT04361799
Title: Perioperative Closed-loop Insulin Delivery Versus Standard Insulin Therapy - a Randomised Controlled Parallel Clinical Trial in Adults With Type 2 Diabetes
Brief Title: Perioperative Closed-loop Glucose Control
Acronym: POP-LOOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POP-LOOP
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Perioperative Hyperglycaemia; Insulin Therapy; Elective Surgery; Closed-Loop Glucose Control; Artificial Pancreas

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Closed-loop insulin therapy (Experimental)
  Interventions: Device: CamAPS
- Standard insulin therapy (Active Comparator)
  Interventions: Drug: Standard insulin therapy

INTERVENTIONS:
Device: CamAPS — Fully automated closed-loop subcutaneous insulin delivery system. A model predictive controller modulates insulin delivery every 10-12 minutes based on interstitial glucose measurements.
  Arms: Closed-loop insulin therapy
Drug: Standard insulin therapy — Standard insulin therapy according to local clinical practice.
  Arms: Standard insulin therapy

SUMMARY:
The prevalence of diabetes and hyperglycaemia in surgical patients is rising and associated with grater complication rates, length of stay and mortality rates. Suboptimal glucose management in the perioperative setting remains a major barrier to optimal surgical care. While there are guidelines to manage perioperative diabetes care, implementation is challenging and inconsistent, in part due to a stretched workforce, involvement of several disciplines and clinical teams and shortcomings in clinical training and knowledge. Closed-loop glucose control represents an emerging diabetes treatment modality that autonomously adjusts insulin delivery according to continuously measured glucose levels. The use of fully automated closed-loop insulin delivery may represent an easy-to-adopt approach for safe and effective perioperative diabetes management.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* The subject is aged 18 years or over
* Diagnosis of type 2 diabetes using standard diagnostic practice (37)
* The subject is planned for an elective abdominal, thoracic or cardiovascular surgery at the University Hospital Bern expected to last ≥2 hours
* The subject requires treatment with subcutaneous insulin as part of the perioperative glucose management
* The subject is literate in German
* The subject is willing to wear study devices 24/7

Exclusion Criteria:

* Physical or psychological condition likely to interfere with the normal conduct of the study and interpretation of the study results as judged by the investigator
* Known or suspected allergy to insulin
* Type 1 diabetes
* Pregnancy, planned pregnancy, or breast feeding
* Medically documented allergy towards the adhesive (glue) of plasters or unable tolerate tape adhesive in the area of sensor placement
* Lack of safe contraception for female participants of childbearing potential for the entire study duration (medically reliable method of contraception are considered oral, injectable, or implantable contraceptives, intrauterine contraceptive devices, or any other methods judged as sufficiently reliable by the investigator in individual cases).
* Serious skin diseases located at places of the body, which potentially are possible to be used for localisation of the glucose sensor
* Illicit drug abuse or prescription drug abuse
* Incapacity to give informed consent
* Droplet/airborne isolation precautions
* Participation in another clinical trial that interferes with the interpretation of the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-09-02 (Actual)

PRIMARY OUTCOMES:
The proportion of time spent in the target glucose range from 5.6 to 10.0 mmol/L based on sensor glucose levels during the time from hospital admission for elective surgery until discharge. | Up to 20 days

SECONDARY OUTCOMES:
Proportion of time spent with sensor glucose values above target (> 10.0 mmol/L) | Up to 20 days
Proportion of time spent with sensor glucose <3.0 mmol/L | Up to 20 days
Average of sensor glucose level | Up to 20 days
Time spent with sensor glucose below target (5.6 mmol/L) | Up to 20 days
Proportion of time spent with sensor glucose levels in significant hyperglycaemia (glucose levels > 20 mmol/L) | Up to 20 days
Standard deviation and coefficient of variation of sensor glucose levels | Up to 20 days
Total daily insulin requirements | Up to 20 days

OTHER OUTCOMES:
Number of severe hypoglycaemic episodes (plasma glucose <2.2 mmol/L) | Up to 20 days
  Safety outcome
Number of clinically significant hyperglycaemic events (>20.0 mmol/L) with ketonaemia (beta-hydroxybutyrate >1.0 mmol/L) | Up to 20 days
  Safety outcome
Post-surgery comorbidity score as assessed using the Clavien Dindo Classification | Up to 20 days
  The Clavien Dindo Classification consists of 7 grades (I, II, IIIa, IIIb, IVa, IVb and V). The higher the grade, the higher the post-operative comorbidity burden.
Length of hospital stay | Up to 20 days
Proportion when closed-loop was active | Up to 20 days
  Utility outcome (will only be assessed in the closed-loop group)

CONTACTS AND LOCATIONS:
Overall Officials: Lia Bally, MD PhD, Principal Investigator — Department of Diabetes, Endocrinology, Nutritional Medicine and Metabolism, Inselspital, Bern University, Unviersity of Bern
Locations (1):
- Department of Diabetes, Endocrinology, Clinical Nutrition and Metabolism, Inselspital, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krutkyte G, Roos J, Schuerch D, Czerlau C, Wilinska ME, Wuethrich PY, Herzig D, Hovorka R, Vogt AP, Gloor B, Bally L. Fully Closed-Loop Insulin Delivery in Patients Undergoing Pancreatic Surgery. Diabetes Technol Ther. 2023 Mar;25(3):206-211. doi: 10.1089/dia.2022.0400. Epub 2022 Dec 14. PMID 36449375
- [Derived] Herzig D, Suhner S, Roos J, Schurch D, Cecchini L, Nakas CT, Weiss S, Kadner A, Kocher GJ, Guensch DP, Wilinska ME, Raabe A, Siebenrock KA, Beldi G, Gloor B, Hovorka R, Vogt AP, Bally L. Perioperative Fully Closed-Loop Insulin Delivery in Patients Undergoing Elective Surgery: An Open-Label, Randomized Controlled Trial. Diabetes Care. 2022 Sep 1;45(9):2076-2083. doi: 10.2337/dc22-0438. PMID 35880252